CLINICAL TRIAL: NCT00019136
Title: TREATMENT OF PATIENTS WITH ADVANCED EPITHELIAL OVARIAN CANCER USING ANTI-CD3 STIMULATED PERIPHERAL BLOOD LYMPHOCYTES TRANSDUCED WITH A GENE ENCODING A CHIMERIC T-CELL RECEPTOR REACTIVE WITH FOLATE BINDING PROTEIN
Brief Title: Gene Therapy and Biological Therapy in Treating Patients With Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064488; NCI-96-C-0011; NCI-T95-0040N; NCT00001494 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2003-12

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — aldesleukin

INTERVENTIONS:
Biological: MOv-gamma chimeric receptor gene
Biological: aldesleukin
Biological: therapeutic allogeneic lymphocytes

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill ovarian cancer cells. Interleukin-2 combined with white blood cells that are gene-modified to recognize and kill ovarian cancer cells may be an effective treatment for recurrent or residual ovarian cancer.

PURPOSE: Phase I trial to study the effectiveness of interleukin-2 plus gene-modified white blood cells in treating patients who have advanced ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical response in patients with advanced ovarian epithelial cancer treated with intravenously administered allogeneic peripheral blood mononuclear cell-stimulated, gene-modified lymphocytes (MOv-PBL).
* Evaluate the ability of intravenously administered MOv-PBL to traffic to sites of ovarian cancer.
* Determine the duration of survival of transduced lymphocytes in the systemic circulation and at the tumor site in these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified by eligibility to receive interleukin-2 (IL-2) (yes vs no).

Patients undergo leukapheresis. The collected peripheral blood lymphocytes (PBLs) are stimulated with allogeneic peripheral blood mononuclear cells (PBMCs) followed by retroviral transduction with antiovarian cancer MOv-gamma chimeric receptor gene (MOv-PBL). MOv-PBL are then reinfused IV over 30-60 minutes followed by IL-2 IV over 15-30 minutes every 12 hours for up to 8 doses (if eligible). This course may be repeated at least once, beginning 2-3 weeks later. Patients receiving allogeneic PBMC-stimulated PBLs receive donor PBMCs subcutaneously at 1 and 8 days after each MOv-PBL infusion instead of IL-2.

Cohorts of 3-6 patients in each stratum receive escalating doses of MOv-PBL until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 10 patients receive MOv-PBL, without IL-2, followed by immunization with donor PBMCs as above.

Patients are followed at 4 and 8 weeks and then periodically for survival.

PROJECTED ACCRUAL: Approximately 13-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent, resected recurrent, or residual ovarian epithelial cancer
* Failed prior standard effective therapy including cisplatin/carboplatin or paclitaxel
* Tumor positive for folate-binding protein by monoclonal antibody MOv18 binding
* Measurable disease by CT scan, MRI, ultrasound, or physical exam OR
* Minimal residual disease on laparotomy, laparoscopy, or peritoneal washings (i.e., disease not evaluable radiologically or on physical exam)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0 or 1

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 9.0 g/dL
* No coagulation disorder

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* Other liver function tests less than 3 times upper limit of normal
* Hepatitis B antigen negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No major cardiovascular illness
* If history of ischemic heart disease, congestive heart failure, or cardiac arrhythmias, not eligible to receive interleukin-2

Pulmonary:

* FEV_1 and DLCO greater than 70% predicted
* No major respiratory illness

Immunologic:

* Must have an intact immune system as evidenced by a positive reaction to Candida albicans, mumps, or tetanus toxoid skin tests on a standard anergy panel
* HIV negative
* No active systemic infection

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 2 weeks since prior biologic therapy

Chemotherapy:

* See Disease Characteristics
* More than 2 weeks since prior chemotherapy

Endocrine therapy:

* More than 2 weeks since prior endocrine therapy
* No concurrent steroids

Radiotherapy:

* More than 2 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* Prior debulking allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-02

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Pinte L, Cunningham A, Trebeden-Negre H, Nikiforow S, Ritz J. Global Perspective on the Development of Genetically Modified Immune Cells for Cancer Therapy. Front Immunol. 2021 Feb 15;11:608485. doi: 10.3389/fimmu.2020.608485. eCollection 2020. PMID 33658994